CLINICAL TRIAL: NCT04071600
Title: Intranasal Neuropeptide Y in Clinical Trial in Level Two Trauma Patients for PTSD and Acute Stress Disorder (ASD)
Brief Title: Intranasal Neuropeptide Y in Clinical Trial in Level Two Trauma Patients for PTSD and Acute Stress Disorder
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New York Medical College (Other)
Collaborators: Westchester Medical Center (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Esther Sabban, Professor, New York Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13038
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute
Keywords: neuropeptide Y; intranasal; biomarkers; anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute; Anxiety Disorders | interventions — Neuropeptide Y

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Type two trauma patients randomly assigned to be administered the vehicle (water) with Kurve intranasal device once and followed for up to 60 days afterwards for development of Acute Stress Disorder and Posttraumatic Stress Disorder.
  Interventions: Other: Placebo
- Neuropeptide Y (Active Comparator): The individuals in this arm will be randomly assigned to be administered intranasal NPY with Kurve intranasal device once and will be followed for at least 60 days afterwards for development of Acute Stress Disorder and Posttraumatic Stress Disorder.
  Interventions: Drug: Neuropeptide Y
- Control (No Intervention): The individuals in this arm will be randomly assigned and treated the same as the other arms but with no intervention.

INTERVENTIONS:
Drug: Neuropeptide Y — Intranasal
  Arms: Neuropeptide Y
Other: Placebo — intranasal
  Other Names: vehicle
  Arms: Placebo

SUMMARY:
Level 2 trauma patients admitted to Westchester Medical Center who consent and meet the inclusion criteria will answer a questionnaire, be tested on Beck Anxiety Index, assessed for vital signs and provide blood and urine samples for biomarker testing. before the intervention.

Part 1 Dose Escalation: Subjects will receive a single infusion NPY or vehicle delivered to the upper nasal cavity with an intranasal device. The administration of intranasal NPY will follow the 3 plus 3 model and Fibonacci dose escalation scheme.

Subjects will be assessed for Acute Stress Disorder (ASD) on the National Stressful Events Survey Acute Stress Disorder Sheet (NSESSS) at 3-7 and at 14-30 days post trauma, At >60 days post trauma to be evaluated with the PTSD Symptom Scale Interview for DSM-5 (PSS-I-5) and given the Beck Anxiety Inventory test.

Part 2 Dose Expansion Cohort: Once the maximal tolerated dose (MTD) is determined, we will follow it by a dose expansion cohort to obtain preliminary evidence of efficacy of intranasal NPY to alter the severity of ASD and inhibit the progression to PTSD and the usefulness of several biomarkers.

DETAILED DESCRIPTION:
Patients admitted to the Westchester Medical Center as a level 2 trauma patient who meet the admission criteria will be asked to join the study and written consent will be obtained. Every patient who consents to participate will fill out a questionnaire of general information including education level, marital status, social support etc. and administered the Beck Anxiety Inventory. They will be asked to collect urine samples until the next morning.

The next morning at about 9-11 AM vital signs will be measured, including standing systolic blood pressure. Blood and the overnight urine samples will be collected for biomarker testing. This will include urinary norepinephrine levels, plasma ACTH and epigenetic changes in the genes for glucocorticoid receptor and norepinephrine transporter.

Subjects will then receive intranasal NPY (GMP-grade) delivered to the upper nasal cavity with an intranasal device from Kurve. We have chosen this device since it appears to be the best delivery system to the upper olfactory region of the nose for delivery to the brain. It has been used most widely, including the earlier clinical trial with intranasal NPY. After the intranasal NPY, patients will be evaluated for potential adverse reactions and vital signs measured at 30 min, 90 min, and every 4 hrs until released from the hospital. 1 and 3 days after the intranasal infusion.

The dose escalation of intranasal NPY will follow the 3 plus 3 model and Fibonacci dose escalation scheme with a starting dose of 9.6mg, selected based on the highest previously studied dose (Sayed et al. 2018). According to this model if no participant has a dose limiting toxicity (DLT), we will proceed to the next dose. If 1/3 has a DLT, 3 additional participants will be enrolled and if more than 1/6 have a DLT the dose escalation will be terminated.

A DLT will be defined as an adverse event or a clinically significant change in vital signs as follows: (1) any serious adverse event experienced at any time during the study that was determined to be at least "possibly" related to the study drug, or (2) a non-serious adverse event rated at least moderate in severity and at least "possibly" related to the study drug, or (3) occurrence of any of the following changes in vital signs with 90 minutes following administration of the NPY: (i) symptomatic hypotension or >20% decrease in systolic blood pressure (SBP) and an absolute SBP < 90; (ii) symptomatic hypertension or >20% increase in SBP and an absolute SBP >170 or diastolic blood pressure (DBP) > 95; (iii) new onset of tachyarrhythmia (defined as a heart rate >100 bpm) or symptomatic bradycardia (heart rate <60 bpm).

Tests for Persistent ASD and Development of PTSD At 3-7 and 14-30 days post trauma, subjects will be asked to fill out the National Stressful Events Survey Acute Stress Disorder Short Scale (NSESSS). After at least 60 days from the trauma they will be given an interview to be evaluated with the PTSD Symptom Scale Interview for DSM-5 (PSS-I-5) as well as the Beck Anxiety Inventory.

Dose escalation cohort After reaching the maximal tolerated dose (MTD) of intranasal NPY or four dose escalation steps without reaching a DLT, we will add a dose escalation cohort. The individuals in this cohort will be randomly assigned to be administered intranasal NPY or vehicle (placebo).

Based on the statistical analysis, we hope to be able to expand to 25-33 individuals per group in order to detect a 15% reduction in incidence of PTSD beyond the influence of the placebo with power of 80%.

Subjects will be tested for: Persistent ASD (NSESS) at days 3-7 and 14-30 after the trauma, PTSD and t 3-7 and 14-30 days post trauma: development of PTSD ( PSS-I-5), > 60 days post trauma); and anxiety (Beck Anxiety Inventory) and compared to groups given no intervention.

The information is expected provide preliminary data on efficacy of intranasal NPY administration to reduce the severity of ASD and attenuate the progression to PTSD. In addition, the results should provide preliminary information on usefulness of several biomarkers to inform on the progression of ASD and PTSD in level 2 trauma patients and on the response to intranasal NPY.

ELIGIBILITY:
Inclusion Criteria:

* Level 2 trauma patients admitted to the trauma floors or trauma ICU at Westchester Medical Center
* Experienced fear at the time of the trauma

Exclusion Criteria:

* Vulnerable populations, such as pregnant women, prisoners, persons with decisional incapacity.
* History of coronary artery disease, heart failure, prior stroke, heart surgery
* Bood pressure >160/90
* Acutely psychotic
* Current diagnosis of anorexia nervosa, bulimia
* Current diagnosis of cancer
* Drug abuse or dependence in the preceding 3 months,
* Any unstable medical condition
* Active suicidal/homicidal ideation
* Cannot speak, read, write and understand English at least at 8th grade level.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 6-9 months
  Dose escalation until treatment emergent adverse effect
Preliminary indication of efficacy of intranasal NPY compared to placebo and no intervention for PTSD | 2-3 years
  Rating for likely PTSD on PSS-I-5 a 20 item interview >60 days after the trauma
Preliminary indication of efficacy of intranasal NPY compared to placebo and no intervention for early Acute Stress Disorder (ASD) | 2-3 years
  Rating on National Stressful Events Survey Acute Stress Disorder Short Form (NSESS) 3-7 days after traum
Preliminary indication of efficacy of intranasal NPY compared to placebo and no intervention for prolonged Acute Stress Disorder (ASD) | 2-3 years
  Rating on National Stressful Events Survey Acute Stress Disorder Short Form (NSESS) 14-30 days after trauma

SECONDARY OUTCOMES:
Preliminary indication of efficacy of intranasal NPY compared to placebo and no intervention for anxiety | 2-3 years
  Scores on Beck Anxiety Inventory (BAI)
Preliminary indication of usefulness of blood pressure to predict development of ASD and PTSD and response to intranasal NPY | 3 years
  Blood pressure measured sitting and standing
Preliminary indication of usefulness of urinary norepinephrine to predict development of ASD and PTSD and usefulness of intranasal NPY | 3 years
  Urinary norepinephrine levels by ELISA
Preliminary indication of usefulness of plasma ACTH to predict development of ASD and PTSD and response to intranasal NPY | 3 years
  Plasma ACTH by ELISA
Preliminary indication of usefulness of epigentic changes in GR and NET genes to predict development of ASD and PTSD and response to intranasal NPY | 3 years
  Methylation of the genes for glucocorticoid receptor (GR) and Norepinephrine Transporter (NET)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Sabban, PhD, Principal Investigator — New York Medical College; Rhea Dornbush, PhD, Principal Investigator — New York Medical College; Yvette Smolin, MD, Principal Investigator — Westchestr Medical Center
Locations (2):
- United States (2):
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center, Valhalla, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sayed S, Van Dam NT, Horn SR, Kautz MM, Parides M, Costi S, Collins KA, Iacoviello B, Iosifescu DV, Mathe AA, Southwick SM, Feder A, Charney DS, Murrough JW. A Randomized Dose-Ranging Study of Neuropeptide Y in Patients with Posttraumatic Stress Disorder. Int J Neuropsychopharmacol. 2018 Jan 1;21(1):3-11. doi: 10.1093/ijnp/pyx109. PMID 29186416
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873